CLINICAL TRIAL: NCT02602223
Title: A Randomized Split-mouth Clinical Trial on Effectiveness of Amnion-Chorion Membranes in Alveolar Ridge Preservation: a Clinical, Radiological, & Morphometric Study
Brief Title: Comparison of Amnion Chorion Membrane vs. Dense Polytetrafluoroethylene Membrane in Ridge Preservation Procedures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Snoasis Medical Products (Industry)
Responsible Party: Principal Investigator, Sivaraman Prakasam, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1207009182
Record Dates: First submitted 2015-11-08; First posted 2015-11-11 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Alveolar Bone Loss; Pathological Conditions, Anatomical
Keywords: Alveolar Ridge Augmentation; Tooth Socket; Guided Tissue Regeneration; Membranes
MeSH Terms: conditions — Alveolar Bone Loss; Pathological Conditions, Anatomical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amnion chorion membrane (Experimental): Amnion chorion membrane will be placed over bone graft after socket preservation on randomly assigned side of the mouth i.e., contra-lateral to the active comparator.
  Interventions: Device: Placing Amnion chorion membrane over grafted site
- d-PTFE membrane (Active Comparator): dense polytetrafluoroethylene membrane will be placed over bone graft after socket preservation on randomly assigned side of the mouth i.e., contra-lateral to the Experimental side
  Interventions: Device: Placing d-PTFE membrane over grafted site

INTERVENTIONS:
Device: Placing Amnion chorion membrane over grafted site — Selected teeth were extracted with minimal trauma to hard and soft tissues. The extraction sites were evaluated to verify presence of intact socket walls. Sockets were thoroughly debrided and a combination of demineralized freeze-dried bone and mineralized freeze-dried bone allograft from a single lot number (Maxxeus, Ohio, U.S.A) was placed in the sockets. Per randomization protocol ACM (BioXclude, Snoasis Medical, Colorado, U.S.A were tucked into the buccal and lingual flaps, which were minimally elevated (2-3mm) and d-PTFE sutures (Osteogenics Medical, Texas, U.S.A) were used to keep membrane in place. Primary closure was not attempted and membranes were intentionally left exposed
  Other Names: BioXclude
  Arms: Amnion chorion membrane
Device: Placing d-PTFE membrane over grafted site — Selected teeth were extracted with minimal trauma to hard and soft tissues. The extraction sites were evaluated to verify presence of intact socket walls. Sockets were thoroughly debrided and a combination of demineralized freeze-dried bone and mineralized freeze-dried bone allograft from a single lot number (Maxxeus, Ohio, U.S.A) was placed in the sockets. Per randomization protocol d-PTFE membranes (Cytoplast, Osteogenics Medical, Texas, U.S.A) were tucked into the buccal and lingual flaps, which were minimally elevated (2-3mm) and d-PTFE sutures (Osteogenics Medical, Texas, U.S.A) were used to keep membrane in place. Primary closure was not attempted and membranes were intentionally left exposed
  Other Names: Cytoplast
  Arms: d-PTFE membrane

SUMMARY:
The purpose of this study is to examine if a biologically active commercially available amnion chorion membrane (ACM) is as effective as the commercially available inert dense polytetrafluoroethylene membrane (D-PTFE) in preserving jaw bone dimensions and whether it provides the added benefit of reducing post-operative discomfort after dental surgery

DETAILED DESCRIPTION:
The purpose of this study is to examine if a biologically active commercially available amnion chorion membrane (ACM) is as effective as the commercially available inert dense polytetrafluoroethylene membrane (D-PTFE) in preserving jaw bone dimensions and whether it provides the added benefit of reducing post-operative discomfort after dental surgery. The hypotheses for the study is that the use of ACM in preservation of bone dimensions in extraction socket will result in greater remaining horizontal and vertical ridge dimension, and reduced postoperative discomfort when compared with D-PTFE in sites where extraction socket will not be closed by advancing the gums. Subjects in need of single rooted teeth extraction on both left and right side of the same jaw will be recruited. Pre-surgical clinical and radiological measurements will be made using dental calipers, stents and reduced cone beam computed tomography (CBCT) three dimensional scans. Involved teeth will be extracted with minimal trauma. Freeze dried bone allograft (bone from human donors) will be used in all extraction sockets. ACM will be used in the one extraction socket and D-PTFE in the other extraction socket without advancing the gums to cover the socket. A Visual Analog Score (VAS), pain scale questionnaire will be given to record the postoperative discomfort and patient will be seen for routine post-operative monitoring as well as research measurements. At 3-months recall postoperatively, clinical measurements and radiographic measurements will be recorded as before. Wound fluid will also be collected at all visits. The sites will be reentered and trephine core (bone sample) will be collected for histomorphometric as well as microtomographic assessment. Statistical analysis will be performed to test the significance using a mixed-model analysis of variance (ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* Subjects needing bilateral non-molar dental extractions in the same arch and consenting to a 2nd surgery for core-biopsy participated in the study. Subjects were required to be within the American Academy of Anesthesiologists (ASA) classifications ASA I or ASA II. Males between 18-75 years and females between 18-50 years of age were screened.

Exclusion Criteria:

* inability or anticipated failure to maintain adequate oral hygiene; evidence of active periodontitis; pregnant or breastfeeding mothers, unstable systemic diseases or with compromised immune system (e.g., uncontrolled diabetes, etc.) or unstable bleeding disorders; active infectious diseases (e.g., hepatitis, tuberculosis, HIV, etc.); mental disabilities that may hinder participation; active immunosuppressive therapy, cancer therapy and/or radiation to the oral cavity within last 6-months; conditions/medications contraindicated for bone regeneration (e.g., methotrexate, steroids, bisphosphonates, cyclosporin-A), and and self-reported tobacco usage (equivalent to >20 cigarettes per day).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sivaraman Prakasam, BDS., MSD., PhD, Principal Investigator — Oregon Health & Science University & Indiana University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening, recruitment and study-related procedures were done at Indiana University School of Dentistry (IUSD) clinics between 9/17/2012 and 7/14/2014
Groups:
- Amnion Chorion Membrane & d-PTFE: Amnion chorion membrane or d-PTFE will be placed over bone graft after socket preservation on randomly assigned side of the mouth i.e., contra-lateral to the active comparator.
  Placing Amnion chorion membrane or d-PTFE over grafted site: Selected teeth were extracted with minimal trauma to hard and soft tissues. The extraction sites were evaluated to verify presence of intact socket walls. Sockets were thoroughly debrided and a combination of demineralized freeze-dried bone and mineralized freeze-dried bone allograft from a single lot number (Maxxeus, Ohio, U.S.A) was placed in the sockets. Per randomization protocol ACM or d-PTFE (BioXclude, Snoasis Medical, Colorado, U.S.A were tucked into the buccal and lingual flaps, which were minimally elevated (2-3mm) and d-PTFE sutures (Osteogenics Medical, Texas, U.S.A) were used to keep membrane in place. Primary closure was not attempted and membranes were intentionally left exposed.
Period: Overall Study
Arm/Group | Amnion Chorion Membrane & d-PTFE
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Amnion Chorion Membrane & d-PTFE
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: Years] | 54.88 [34 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 9
Total Number of sites (maxilla vs Mandible) [Number; unit: Sites] — Number of sites in maxilla that received either ACM or d-PTFE
  Sites
    Total | 22
    Maxilla | 14
    Mandible | 8
Number of participants with multiple study sites [Number; unit: participants] — Number of participants who received either single vs multiple bilateral sites
  participants
    Single paired study sites | 7
    Multiple (two) paired study sites | 2

OUTCOME MEASURES:

1. Primary Outcome: Amount of Preservation of Alveolar Ridge Dimensions i.e..,Clinical Horizontal Ridge Width Change in Millimeter as Result of Ridge Preservation Procedures
Description: A radiographic stent will be fabricated with reproducible access holes ≈5 mm apical to the mid-facial and mid-lingual gingival margin of the teeth to be extracted. On day of surgery, a calibrated examiner masked to treatment allocation, will record initial clinical bucco-lingual (iCBL) ridge measurements in millimeters (mm), through the access holes in the stent, using calipers. Approximately 3.5(±0.5)-months post extractions, the calibrated examiner masked to treatment allocation, will record the final clinical bucco-lingual (fCBL) ridge measurements in mm using the calipers as described earlier. The difference between fCBL and iCBL will be calculated as change in clinical horizontal ridge width dimensions in mm (cΔHD).
Time Frame: 3-4 months
Population: change in clinical horizontal ridge width dimensions in mm - cΔHD
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Sites
Arm/Group | Amnion Chorion Membrane | d-PTFE Membrane
Number analyzed (Participants) | 9 | 9
Number analyzed (Sites) | 11 | 11
millimeters | 2.54 (1.29) | 2.72 (1.01)

2. Primary Outcome: Evaluation of Preservation of Ridge Quality Through Microtomographic Analysis for Microarchitectural Parameters Expressed as Percentages.
Description: Approximately 3-months post extractions, a 2.5x10mm core of bone will be removed from the center of the residual ridge using a 2.5mm inner-diameter trephine bur. Cores will be immediately placed into 10%-formalin. A high-resolution microtomographic scanner will be used and images will be scanned at a voxel size of 8µm3. Moist bone cores will be wrapped in paraffin and scanned in air. Cores will be rotated in 0.7 degree increments with 450milli second time exposition. A 0.5m aluminum filter will be used to remove image noise. After scanning, 3D microstructural image data will be reconstructed using software. Structural indices will be calculated using a software. The micro-architectural variables; bone volume density (BV/TV), and bone surface density (BS/BV); will be quantified and reported as percentages.
Time Frame: 3-4 month
Population: The micro-architectural variable; bone volume density (BV/TV),was quantified and is reported as percentages.
Measure: Mean (Standard Deviation); unit: Percentage of BV/TV
Arm/Group | Amnion Chorion Membrane | d-PTFE Membrane
Number analyzed (Participants) | 9 | 9
Percentage of BV/TV | 51.74 (17.13) | 37.31 (11.93)

3. Primary Outcome: Evaluation of Preservation of Ridge Quality Through Histological Analysis for Microarchitectural Parameters Expressed as Percentages.
Description: Approximately 3.5(±0.5)-months post extractions, a 2.5x10mm core of bone will be removed from the center of the residual ridge using a 2.5mm inner-diameter trephine bur. Cores will be immediately placed into 10%-formalin. Cores will be process and embedded in polymethylmethacrylate and sectioned to 5μm thickness and sections will be stained with Goldener's Trichrome. With the Goldener's trichrome, mineralized bone appears as green or blue regions, osteoid appears orange-red, nuclei appears blue-grey and graft remnants appear grey. Additional differentiation between graft and new bone will be achieved by morphologically assessing each sample individually. A slide scanner will be used to image the sample (20x magnification), and a software program will be used for the histomorphometric analysis, to quantify the amount of total mineralized bone, new bone / osteoid, soft tissue, and residual graft remnants in percentages .
Time Frame: 3-4 months
Population: New bone/osteoid Percentages
Measure: Mean (Standard Deviation); unit: Percentage of New bone
Arm/Group | Amnion Chorion Membrane | d-PTFE Membrane
Number analyzed (Participants) | 9 | 9
Percentage of New bone | 8.31 (8.20) | 3.50 (3.59)

4. Primary Outcome: Post Operative Pain
Description: A visual Analog score (VAS) pain scale form (scale of 1 to 10) will be provided with instructions to record pain levels on both surgical sites every day for 2-weeks post-surgery. VAS score of 10 indicates highest level of pain and 0 indicates no pain. Subjects will also asked to log any pain medications taken in that 2-week period. Subjects will be seen at 1&2 weeks for post-operative evaluation and VAS forms will be collected. Data will be reported as Average VAS score.
Time Frame: 0-2 weeks
Population: VAS score at 24 hours post operative
Measure: Mean (Standard Deviation); unit: Units on a scale of 10
Arm/Group | Amnion Chorion Membrane | d-PTFE Membrane
Number analyzed (Participants) | 9 | 9
Units on a scale of 10 | 1.82 (1.57) | 4.09 (2.7)

5. Primary Outcome: Amount of Preservation of Alveolar Ridge Dimensions Following Ridge Preservation Procedures i.e., Horizontal Ridge Width Height Change in Millimeters as Assessed Through Analysis of CBCT Scans.
Description: Radiographic stent with radiopaque reference plane (RRP) will be used to obtain pre-extraction CBCT scans. Approximately 3-months post extractions, a second CBCT will be taken. Radiographic Analyses will be done using radiographic image analysis software by a calibrated examiner. The initial relative crest (iRC) reference point will be determined. The buccal and lingual crests at the central plane of site will be marked and distances from this crest to RRP will be measured in mm. The average distance of the buccal crest height and the lingual crest height will be calculated and that value will be used to determine the iRC for that site. Initial Bucco-lingual (iRBL) measurements will be recorded at 1 mm, 3 mm and 7 mm from iRC in all five planes. The final bucco-lingual (fRBL) measurements will be recorded on the second CBCT, using the same method as described before and using the iRC reference. Differences between iRBL and the fRBL reflect change in horizontal ridge width (RΔHD).
Time Frame: 3-4 months
Population: Change in horizontal ridge width (RΔHD).
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Amnion Chorion Membrane | d-PTFE Membrane
Number analyzed (Participants) | 9 | 9
millimeters | 1.33 (0.72) | 2.53 (3.34)

6. Primary Outcome: Amount of Preservation of Alveolar Ridge Dimensions Following Ridge Preservation Procedures i.e., Vertical Ridge Height Change in Millimeters as Assessed Through Analysis of CBCT Scans.
Description: Radiographic stent with a radiopaque reference plane (RRP) will be used to obtain pre-extraction CBCT scans. Approximately 3.5(±0.5)-months post extractions, a second CBCT will be taken. Radiographic Analyses will be done using radiographic image analysis software by a calibrated examiner. Initial relative crest iRC will be determined as described above from the initial CBCT. In the second CBCT, vertical distance from the iRC from initial CBCT will be used to recreate the iRC. New relative crest will be determined for each of the three planes (nRC) as above. The difference between iRC and nRC indicates change in vertical dimension at each plane (RΔVD) i.e., iRC - nRC = (RΔVD). Positive (RΔVD) values indicate relative loss of crestal bone height and negative (RΔVD) values indicate relative gain of crestal bone height.
Time Frame: 3-4 months
Population: Change in vertical dimension at each plane (RΔVD) i.e., iRC - nRC = (RΔVD). Positive (RΔVD) values indicate relative loss of crestal bone height and negative (RΔVD) values indicate relative gain of crestal bone height.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Amnion Chorion Membrane | d-PTFE Membrane
Number analyzed (Participants) | 9 | 9
millimeters | -0.24 (0.91) | 1.18 (2.22)

ADVERSE EVENTS:
Arm/Group | Amnion Chorion Membrane | d-PTFE Membrane
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
Small Sample size, but expanding study not justified through post hoc analysis. Crossover effects due to split mouth study design potentially indirect and possibly only minimal due to biological infeasibility of cross over effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No